CLINICAL TRIAL: NCT06271161
Title: The Effect of Pharyngeal Cooling Applications on Postoperative Throat Pain and Nausea Vomiting
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Assisstant Professor, Selcuk University
Other Study IDs: F002
Record Dates: First submitted 2024-01-25; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Throat, Sore; Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Pharyngitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to to evaluate the effects of a throat pack soaked with saline at +4 ºC on postoperative throat pain (POTP) and postoperative nausea and vomiting (PONV) in dental surgical procedures performed under general anesthesia. The main questions it aims to answer are: 1. How long can we keep the pharyngeal mucosa cold using tampons and cold wash solutions? 2. Does cooling the pharyngeal mucosa reduce the incidence of postoperative sore throat and nausea and vomiting?

DETAILED DESCRIPTION:
The study included 84 ASA I - II patients, over 18 years of age, who would undergo outpatient surgery under general anesthesia in the operating room of Selçuk University Faculty of Dentistry. Apfel score was used to classify patients according to PONV risk. Patients with Apfel scores of 0, 1 and 2 were included in the study. Patients with a history of difficult intubation, patients who could not be intubated at the first attempt, patients with bleeding disorders, motion sickness, malignancy, and patients who had an upper respiratory tract infection in the last 2 weeks were excluded from the study.

The patients were not prescribed any analgesics or anxiolytics before surgery. Pulse oximetry (SpO2), electrocardiogram (ECG), non-invasive blood pressure and end-tidal CO2 pressure (PETCO2) and nasopharyngeal temperature measurement (T), which are standard monitoring methods in general anesthesia applications, were applied to all patients and the values were recorded every 5 minutes. Each patient was administered IV cannulation over the right hand and 1 mg/kg intravenous methylprednisolone and 40 mg pantoprozole were administered before surgery. Anesthesia was induced with 3 mg/kg iv sodium thiopental, 0.6 mg/kg iv rocuronium bromide and 1-1.5 mcg/kg iv fentanyl, and was maintained with 2% sevoflurane in 50% N2O/50% O2. All patients were given appropriate head and neck position before surgery, after nasal intubation with an endotracheal tube (ETT) with lubricating gel applied to the cuff, with the help of a videolaryngoscope. ETT cuff pressure was kept within the range of 20-30 cm H2O with the help of a manometer (VBM, Sultz, Germany) throughout the surgery. The patient's body temperature was monitored by placing a reusable temperature probe into the nasopharynx and recorded during the operation. A throat tampon made of 20x10 cm diameter gauze soaked in saline at +4 ºC was gently placed into the oropharynx by the anesthetist and surgical procedures were initiated.

Demographic data of the patients included in the study such as age, gender, weight, Apfel scores, total doses of opioid drugs used in anesthesia, anesthesia-related data such as ASA score, endotracheal tube diameter, and surgical procedure-related data such as surgical time, surgical procedure, and amount of bleeding were recorded.

During the surgery, the operating room temperature was kept between 22 ºC and 24 ºC. The amount of saline at +4 ºC used to wash the oral cavity during surgical procedures was recorded. At the conclusion of the surgical procedures, the neuromuscular blockade was reversed and the tampon was gently removed by the same anesthesiologist before extubation. All patients were administered IV 50 mg Dexketoprofen just before waking up from general anesthesia.

All patients in the study were extubated and taken to the recovery room. Nausea, vomiting, and sore throat were recorded at the 5th, 10th, and 30th minutes, and at the 1st, 2nd, and 6th hours postoperatively by a surgical assistant who was blinded to the study. IV 20 mg metoclorpamide was used as rescue antiemetic. For pain scores higher than POBA 4, 75 mg tramadol in 100 ml 0.9% saline was administered as a 10-minute IV infusion. Analgesic and antiemetic drug use was recorded as present or absent. All patients were discharged on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* > 18 year old
* ASA I-II
* Apfel Score<2

Exclusion Criteria:

* Clinical diagnosis of motion sickness
* Clinical diagnosis of malignancy
* Clinical diagnosis of upper respiratory tract infection in last 2 weeks
* Clinical diagnosis of any bleeding disorders
* Patient that couldn't be intubated at first attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 84 patients who were older than 18 years of age and had ASA (American Society of Anesthesiologists) physical status classification I - II, who underwent outpatient dental surgical procedures under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative sore throat and noise vomiting was investigated in dental surgery involving the application of cooling to the pharyngeal area, particularly when a throat pack was used. | 1 month
  The incidence of postoperative throat pain (POTP) was recorded with the following 100 mm VAS scale: 0, no POTP; 1-3, mild POTP (complaining of throat pain only when asked); 4-7, moderate POTP (complaining of throat pain spontaneously); and 8-10, severe POTP (presence of voice change or hoarseness accompanying throat pain). Additionally, the incidence of postoperative nausea and vomiting (PONV) was assessed at the 5th, 10th, and 30th minutes, as well as at the 1st, 2nd, and 6th hours, using the following Myles's simplified PONV impact scale (score > 0 is regarded as the occurrence of PONV, vomited or dry-retching (0-3 score) and nausea (0-3 score) ,with higher scores indicating being more severe.

SECONDARY OUTCOMES:
Intraoperative change in nasopharyngeal temperature from baseline (ºC ), intraoperative opioid usage (mcg), postoperative analgesic usage (mg),antiemetic usage(mg) and any adverse events due to throat pack were recorded. | 1 month
  During the surgery, the patient's nasopharyngeal temperature(ºC ), total doses of opioid drugs used (mcg), analgesic and antiemetic drug use (yes/no) in the postoperative recovery room, and the presence/absence of any undesirable events related to the throat pack were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: FUNDA ARUN, Ass. Prof., Principal Investigator — Selcuk University Faculty of Dentistry
Locations (1):
- Funda Arun, Selçuklu, Konya, Turkey (Türkiye)